CLINICAL TRIAL: NCT01049750
Title: Prevalence and Risk Factors of Erectile Dysfunction in Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Professor, University of Pavia
Other Study IDs: 20090001127; P-20090002836 (Registry Identifier: 20090002304)
Record Dates: First submitted 2010-01-11; First posted 2010-01-14 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetic Patients; Erectile Dysfunction
Keywords: type 2 diabetes mellitus; male; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- type 2 diabetic patients: males; type 2 diabetic patients
  Interventions: Other: type 2 diabetic patients

INTERVENTIONS:
Other: type 2 diabetic patients — males; type 2 diabetic patients

SUMMARY:
The investigators evaluated 250 male, type 2 diabetic patients, aged 18-80 years. They will undergo IIEF (International Index of Erectile Function), SAS of Zung (self-rating anxiety state)and SDS of Zung (self-rating depression scale)questionnaires. The investigators will evaluate anthropometric and biochemical parameters, dysautonomic function index, IMT (Intima Media Thickness) index, and fundus oculi examen. Furthermore, the investigators will perform MNSI (Michigan Neuropathy Screening Instrument) and NDS (Neuropathy Disability Score)questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus

Exclusion Criteria:

* type 1 diabetes mellitus
* < 18 years old
* anatomic abnormalities of the penis
* patients taking erectile dysfunction therapy at the moment of the enrollment

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: males with type 2 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2009-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of erectile dysfunction | Baseline (time 0); 3 months; 6 months
Description of erectile disfunction markers | Baseline (time 0); 3 months; 6 months
Evaluation of diabetic neuropathy in patients with erectile dysfunction | Baseline (time 0); 3 months; 6 months

SECONDARY OUTCOMES:
Metalloproteinases 2 and 9 | Baseline (time 0); 3 months; 6 months
Insulin-sensitivity index (HOMA index) | Baseline (time 0); 3 months; 6 months
Glycemic control | Baseline (time 0); 3 months; 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, Principal Investigator — University of Pavia - Fondazione IRCCS Policlinico San Matteo - Pavia
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Result] Derosa G, Tinelli C, D'Angelo A, Ferrara G, Bonaventura A, Bianchi L, Romano D, Fogari E, Maffioli P. Glyco-metabolic profile among type 2 diabetic patients with erectile dysfunction. Endocr J. 2012;59(7):611-9. doi: 10.1507/endocrj.ej12-0117. Epub 2012 May 26. PMID 22572549
- [Result] Derosa G, Romano D, Tinelli C, D'Angelo A, Maffioli P. Prevalence and associations of erectile dysfunction in a sample of Italian males with type 2 diabetes. Diabetes Res Clin Pract. 2015 May;108(2):329-35. doi: 10.1016/j.diabres.2015.01.037. Epub 2015 Feb 7. PMID 25747572